CLINICAL TRIAL: NCT04035863
Title: EVALUATION OF THE SENSORY-MOTOR RESPONSE IN PATIENTS WITH MYELOMENINGOCELE FOLLOWING TREATMENT WITH PHOTOBIOMODULATION
Brief Title: Effects of Photobiomodulation on Superficial Sensitivity and Muscle Activity of Individuals With Myelomeningocele
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MieloTamiris
Record Dates: First submitted 2019-07-24; First posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Myelomeningocele Without Hydrocephalus; Sensory Defect; Motor Activity
MeSH Terms: conditions — Motor Activity | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PBM + physiotherapy exercises (Experimental): will be submitted to active PBM and physiotherapeutic exercises.
  For irradiation, the individuals will be positioned comfortably in lateral decubitus on the examining table. Three points will be irradiated at the lesion level with a wavelength of 808 nm, 25 J per point for 12 sessions. The same laser device (Laser DMC Therapy EC).
  Physical therapy will occur twice per week after PBM for six weeks. Static balance exercises will be performed with the feet together and tandem on a variety of different surfaces (hard surface, foam rubber and carpets with different textures) and sensory inputs (eyes open and closed). Dynamic balance exercises will involve walking forward and backward on firm and foam surfaces and circumventing obstacles. Muscle strengthening exercises, squatting and changing postural positions will also be performed. All activities will be in the form of play to maintain the children's interest
  Interventions: Device: Low level laser therapy
- SHAM PBM + physiotherapy exercises (Sham Comparator): will be submitted to sham PBM and physiotherapeutic exercises.
  For irradiation sham, the individuals will be positioned comfortably in lateral decubitus on the examining table. The same laser device (Laser DMC Therapy EC) will be used but the device will emit sound but not light.
  Physical therapy will occur twice per week after PBM for six weeks. Static balance exercises will be performed with the feet together and tandem on a variety of different surfaces (hard surface, foam rubber and carpets with different textures) and sensory inputs (eyes open and closed). Dynamic balance exercises will involve walking forward and backward on firm and foam surfaces and circumventing obstacles. Muscle strengthening exercises, squatting and changing postural positions will also be performed. All activities will be in the form of play to maintain the children's interest
  Interventions: Device: Low level laser therapy

INTERVENTIONS:
Device: Low level laser therapy — For the PBM protocol, articles of interest were identified through analyses of titles and abstracts. Articles addressing PBM in experimental models or clinical trials of spinal cord injuries were included and articles not pertinent to the proposed study were excluded. Next, the selected articles were analyzed and used for the creation of an initial protocol (Table 1).
  For irradiation, the individuals will be positioned comfortably in lateral decubitus on the examining table. Three points will be irradiated above the lesion level, which will be located using an imaging exam brought by the guardian on the day of the evaluation. After determining the lesion level, palpation of the transverse processes of the vertebrae will be performed. The same laser device (Laser DMC Therapy EC) will be used for both groups. For the placebo group, the device will emit sound but not light.

SUMMARY:
Myelomeningocele is a neural tube defect that occurs between the third and fourth week of gestation. Functional impairment occurs due to dysplasia of the nerve roots, which can lead to flaccid paralysis and sensory-motor dysfunction below the level of the lesion. Although advances in the multidisciplinary treatment of myelomeningocele have led to functional improvements in affected children, novel therapeutic modalities, such as photobiomodulation (PBM), could be a promising complement to treatment. Objective: Evaluate the effectiveness of PBM combined with physiotherapeutic exercises on the sensory-motor response in individuals with myelomeningocele at the lower lumbar and sacral level. Participants will be recruited from the Integrated Health Clinic of University Nove de Julho and randomized into two groups: Grupo 1 - treatment with PBM at a wavelength of 808 nm + physical therapy; Grupo 2 - sham PBM + physical therapy. Evaluations will involve electromyography of the gastrocnemius, tibialis anterior and rectus femoris muscles of both lower limbs. Balance will be evaluated using the Pediatric Balance Scale. The sensory evaluation will be performed using the Semmes-Weinstein monofilament kit (Smiles®). BDNF levels will be determined using ELISA. The data will be analyzed with the aid of GraphPad PRISM version 7.0. The Kolmogorov-Smirnov test will be used to determine the normality of the data. Variables that fit the Gaussian curve will be expressed as mean and standard deviation values. The t-test will be used for the comparisons between groups, with the level of significance set to 95% (p < 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Age 5 to 16 years;
* diagnosis of myelomeningocele on the lower lumbar and sacral level;
* community ambulator;
* score above the cutoff point for age on the Mini Mental State Examination.

Exclusion Criteria:

* Cognitive impairment that compromises the ability to communicate and answer the questions that will be posed;
* allergy to latex; - manifestations secondary to MMC, such as hydrocephalus;
* congenital club foot; neuromuscular scoliosis;
* subluxation or luxation of hip and knee;
* other disease of the central nervous system, neoplasms, heart failure, renal, respiratory, hepatic.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2019-09-02 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-05-03 (Estimated)

PRIMARY OUTCOMES:
Assessment of muscle activity | 10 minutes
  Electromyography (EMG) will be performed with the EMG System®. The participants will be placed on an examining table and the skin will be cleaned with tissues soaked in alcohol for the placement of the markers. Disposable self-adhesive Ag/AgCl surface electrodes (Noraxon) measuring 10 mm in diameter will be attached to the belly of the lateral gastrocnemius, tibialis anterior and rectus femoris muscles on both lower limbs to capture the EMG signals. A reference electrode will be placed on the left wrist of the volunteers to impede interference of external noise
Sensory evaluation - monofilaments | 10 minutes
  The sensory evaluation will be performed using the Semmes-Weinstein kit (Smiles®), which is a set of six nylon monofilaments of the same length that exert force on the specific area tested. Each monofilament has a different color and diameter: green (0.05 g), blue (0.2 g), violet (2 g), red (4 g), orang (10 g) and magenta (300 g). The score ranges from seven (green monofilament) to 1 (magenta monofilament). The test will be performed on the following dermatomes: L1, L2, L4, L5, S1, S2 and S3.

SECONDARY OUTCOMES:
Evaluation of balance | 10 minutos
  Balance will be evaluated using the Pediatric Balance Scale, which consists of 14 items scored from 0 to 4 points. The maximum score is 56, with higher scores denoting better balance.
Analysis expression of brain-derived neurotrophic factor (BDNF) | 10 minutes
  BDNF be quantified in saliva samples from the participants using ELISA MAX HUMAN kits (BioLegend), which contain capture and detection antibodies for the precise quantification of each cytokine. All kits will be used following the manufacturer's instructions. The optical density of the samples will be measured in a spectrophotometer at 450 nm.
  Collection of saliva
Analysis expression Interleukin-10 (IL-10) | 10 minutes
  IL-10 will be quantified in saliva samples from the participants using ELISA MAX HUMAN kits (BioLegend), which contain capture and detection antibodies for the precise quantification of each cytokine. All kits will be used following the manufacturer's instructions. The optical density of the samples will be measured in a spectrophotometer at 450 nm.